CLINICAL TRIAL: NCT05584904
Title: A Short Segment of a Single Dry EEG Electrode Allows the Digestive Endoscopy and Operating Theater Staff the Estimation of the Level of Anesthesia During Colonoscopy Sedation
Brief Title: A Single Dry EEG Electrode Allows to Estimate of the Level of Anesthesia During Colonoscopy Sedation.
Status: Completed | Type: Observational
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Collaborators: Auxilium Vitae Volterra (Other)
Responsible Party: Principal Investigator, Alessandro Tani, Head of perioperative medicine and pain therapy Volterra Hospital, Azienda USL Toscana Nord Ovest
Other Study IDs: AUSLNordOvest
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia; Adverse Effect
Keywords: raw EEG, colonoscopy sedation
MeSH Terms: interventions — Nurses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: volunteer anesthesiologists and nurses — 18 not expert in electroencephalography digestive endoscopy and operating room nurses, and 8 anesthesiologists interpreting EEGs obtained with a single electrode EEG

SUMMARY:
We asked to a staff of digestive endoscopy and of the operating room to interpret the EEG traces obtained from a single dry electrode device to estimate the level of anesthesia during colonoscopy. They are required to produce a rank value (1 to 3) proportional to the anesthesia level. The rank values of anesthesia evaluated through the EEG traces will be correlated to the typically used "bispectral index" values simultaneously acquired. The expected efficacy of a low-cost single dry-electrode EEG would allow the monitoring of the level of anesthesia during non operating room procedures such as colonoscopy.

DETAILED DESCRIPTION:
Monitoring of the level of anesthesia has two primary functions: to reduce the incidence of awareness during operation and to avoid too deep anesthesia that is associated with increased risks of mortality and postoperative cognitive impairment. This monitoring can be performed by processed EEG such as "Bispectral Index" that provides a simple interpretation numerical value proportional to the anesthesia level. Nevertheless, "Bispectral index" requires specific tools and disposable material that increases costs for non operating room procedure. Colonoscopy is a non operating room procedure typically performed without or with light sedation, less frequently requires deep sedation. The latter is performed by using Propofol a drug that has a low therapeutic index and might be associated with adverse effects such as respiratory depression, aspiration related to loss of airway reflexes and hypotension. The aim of the present study is to evaluate the reliable interpretation of the raw EEG traces by a staff of digestive endoscopy and operating room for monitoring the level of sedation during non operative room anesthesia to avoid adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* anesthesiologists and nursing staff of the operating room

Exclusion Criteria:

* specific knowledge of electroencephalography

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All the anesthesiologists and nursing staff of the digestive endoscopy and operating room of the Volterra Hospital
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Single dry channel EEG for the monitoring of the level of anesthesia in non-operating room. | two hours
  A staff of digestive endoscopy and operating room after attending a brief course of EEG specifically direct to anesthesia level interpretation, were asked to classify the raw EEG trace obtained with a sigle dry electrode device in 3 levels (1 to 3) according to the following category:
  1 deep sedation, , 2 intermediate state, 3 light sedation or awake according to the BIS level and and coherent with clinical conditions.
  We correlate staff scores produced by classifing the EEG trace with the number automatically and simultaneously produced by the "bispectral index" tool for the measurement of the level of anesthesia.
  The reliability of raw single dry electrode EEG trace, might allow to assist low-cost device for non operating room anesthesia such as for colonoscopy sedation.

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Maria Maddalena Hospital, Volterra, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No
the modalities of this option have not yet been decided

REFERENCES:
- [Background] Barnard JP, Bennett C, Voss LJ, Sleigh JW. Can anaesthetists be taught to interpret the effects of general anaesthesia on the electroencephalogram? Comparison of performance with the BIS and spectral entropy. Br J Anaesth. 2007 Oct;99(4):532-7. doi: 10.1093/bja/aem198. Epub 2007 Jul 24. PMID 17652076